CLINICAL TRIAL: NCT01744496
Title: A Multicenter, Multinational, Double-Blind, Placebo-Controlled, 2-Arm Study to Evaluate the Efficacy of Rotigotine on Parkinson's Disease-Associated Pain
Brief Title: Study to Evaluate the Efficacy of Rotigotine on Parkinson's Disease-Associated Pain
Acronym: DOLORES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB BIOSCIENCES GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PD0004; 2012-002608-42 (EudraCT Number)
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Advanced Idiopathic Parkinson's Disease
Keywords: Parkinson's Disease; Rotigotine; Chronic Pain; Nonmotor symptoms
MeSH Terms: conditions — Parkinson Disease; Chronic Pain | interventions — rotigotine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotigotine (Experimental): Rotigotine Transdermal Patches
  Interventions: Drug: Rotigotine
- Placebo (Placebo Comparator): Placebo Transdermal Patches
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rotigotine — Patches will contain 4 mg / 24 h (20 cm^2), 6 mg/ 24 h (30 cm^2), or 8 mg /24 h (40 cm^2) of Rotigotine. Application of study medication starts at the Baseline Visit. Rotigotine will be administered once daily starting at 4 mg / 24 h. Doses will then be up-titrated in weekly increments of 2 mg / 24 h until optimal or maximum dose (16 mg / 24 h) is reached and the Maintenance Period can be started. The duration of the Titration Period will vary from 1 to 7 weeks ± 3 days. The Maintenance Period will last 12 weeks ± 5 days. Thereafter, during the De-escalation Period, the dose of study medication will be decreased by 2 mg / 24 h every other day. The De-escalation Period may last up to 12 days.
  Other Names: (6S)-6-propyl-[2 (2 thienyl)ethyl]amino-5,6,7,8-tetrahydro-1-naphthalenol
  Arms: Rotigotine
Drug: Placebo — Placebo patches match the size of active patches 20 cm^2, 30 cm^2, or 40 cm^2 and will contain Placebo. Application of Placebo patches starts at the Baseline Visit. Placebo patches will be administered once daily starting with the equivalent of 4 mg / 24 h. Doses will then be up-titrated in weekly equivalents to 2 mg / 24 h until either optimal dose or maximum dose is reached. The maximum dose is the equivalent to 16 mg / 24 h. The duration of the Titration Period will vary from 1 to 7 weeks. The Maintenance Period will last 12 weeks ± 5 days. During the De-escalation Period, the dose of Placebo will be decreased by the equivalent to 2 mg / 24 h every other day. The De-escalation Period may last up to 12 days.
  Arms: Placebo

SUMMARY:
This trial is being conducted to compare the impact of Rotigotine and Placebo on Chronic Pain associated with Parkinson's Disease among patients with advanced stages of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient has advanced idiopathic Parkinson's Disease associated chronic pain assessed by a Likert Pain Scale
* Patient is taking Levodopa with a stable daily dose of at least 200 mg for at least 21 days prior to start
* Hoehn and Yahr stage score of II to IV
* Mini-Mental State Examination (MMSE) score ≥ 25
* If an antidepressant drug is taken, the dose must be stable for at least 21 days

Exclusion Criteria:

* Therapy with a Dopamine Agonist within 21 days prior to start
* Discontinuation from previous Dopamine Agonist Therapy due to lack of efficacy
* Therapy with Dopamine-modulating substances 21 days prior to start
* Therapy with analgesics for the treatment for pain, unless the dose has been stable
* Chronic alcohol or drug abuse
* Medical or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the patient's ability to participate in this study
* Hypersensitivity to any components of the Investigational Medicinal Product (IMP) or comparative drugs
* Atypical Parkinson's Disease Syndrome due to drugs
* History of deep brain stimulation
* Significant skin disease that would make transdermal drug use inappropriate
* Electroconvulsive therapy within 12 weeks prior to start
* Evidence of an Impulse Control Disorder
* Previous diagnosis of severe Restless Legs Syndrome
* Chronic Migraine
* Severe Depression
* Symptomatic Orthostatic Hypotension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (16):
- United States (10):
  - 2113, Gilbert, Arizona
  - 2120, Sunnyvale, California
  - 2109, Tampa, Florida
  - 2107, Chicago, Illinois
  - 2102, Lexington, Kentucky
  - 2118, Advance, North Carolina
  - 2117, Cincinnati, Ohio
  - 2103, Tulsa, Oklahoma
  - 2101, Roanoke, Virginia
  - 2104, Milwaukee, Wisconsin
- 1204, Gera, Germany
- Poland (3):
  - 1607, Gdansk
  - 1603, Krakow
  - 1609, Olsztyn
- Slovakia (2):
  - 1804, Bratislava
  - 1805, Dubnica nad Váhom

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Europe and USA. Recruitment was planned to continue until approximately 64 patients were randomized in the study. Subjects were randomized in a 1:1 ratio to either Rotigotine or Placebo. To achieve this, approximately 28 investigational sites were planned to participate in this hypothesis-generating pilot study.
Pre-assignment Details: The Participant Flow population refers to the Randomized Set (RS). The RS includes all subjects who were randomized.
Groups:
- Placebo: Placebo Transdermal Patches
  Placebo: Placebo patches matched the size of active patches 20 cm^2, 30 cm^2, or 40 cm^2 and contained Placebo. Application of Placebo patches started at the Baseline Visit. Placebo patches were administered once daily starting with the equivalent of 4 mg / 24 h. Doses were then up-titrated in weekly equivalents to 2 mg / 24 h until either optimal dose or maximum dose was reached. The maximum dose was the equivalent to 16 mg / 24 h. The duration of the Titration Period varied from 1 to 7 weeks. The Maintenance Period lasted 12 weeks ± 5 days. During the De-Escalation Period, the dose of Placebo will be decreased by the equivalent to 2 mg / 24 h every other day. The De-Escalation Period might have lasted up to 12 days.
- Rotigotine: Rotigotine Transdermal Patches
  Rotigotine: Patches contained 4 mg / 24 h (20 cm^2), 6 mg/ 24 h (30 cm^2), or 8 mg /24 h (40 cm^2) of Rotigotine. Application of study medication started at the Baseline Visit. Rotigotine was administered once daily starting at 4 mg / 24 h. Doses were then up-titrated in weekly increments of 2 mg / 24 h until optimal or maximum dose (16 mg / 24 h) was reached and the Maintenance Period could be started. The duration of the Titration Period varied from 1 to 7 weeks ± 3 days. The Maintenance Period lasted 12 weeks ± 5 days. Thereafter, during the De-Escalation Period, the dose of study medication was decreased by 2 mg / 24 h every other day. The De-Escalation Period might have lasted up to 12 days.
Period: Titration Period
Arm/Group | Placebo | Rotigotine
Started | 33 | 35
Completed | 31 | 33
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Personal reasons | 0 | 1
Period: Maintenance Period
Arm/Group | Placebo | Rotigotine
Started | 31 | 33
Completed | 27 | 29
Not Completed | 4 | 4
Not completed — Adverse Event | 1 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Subject left town | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population refers to the Safety Set (SS). The SS includes all randomized subjects who received at least 1 dose of study medication.
Groups:
- Placebo: Placebo Transdermal Patches
  Placebo: Placebo patches matched the size of active patches 20 cm^2, 30 cm^2, or 40 cm^2 and contained Placebo. Application of Placebo patches started at the Baseline Visit. Placebo patches were administered once daily starting with the equivalent of 4 mg / 24 h. Doses were then up-titrated in weekly equivalents to 2 mg / 24 h until either optimal dose or maximum dose was reached. The maximum dose was the equivalent to 16 mg / 24 h. The duration of the Titration Period varied from 1 to 7 weeks. The Maintenance Period lasted 12 weeks ± 5 days. During the De-Escalation Period, the dose of Placebo was decreased by the equivalent to 2 mg / 24 h every other day. The De-Escalation Period might have lasted up to 12 days.
- Total: Total of all reporting groups
Arm/Group | Placebo | Rotigotine | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 18 | 23 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (13.8) | 66.5 (11.9) | 65.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 17 | 19 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian / Alaskan native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Black | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  White | 32 | 35 | 67
  Other / mixed | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilograms] | 80.15 (20.00) | 77.80 (13.71) | 78.94 (16.97)
Height [Mean (Standard Deviation); unit: centimeters] | 167.17 (9.92) | 168.63 (9.87) | 167.92 (9.85)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per squaremeter] | 28.54 (6.21) | 27.42 (4.74) | 27.96 (5.49)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to the End of the Maintenance Period in Pain Severity Assessed Using an 11-point Likert Pain Scale
Description: An 11-Point Likert Scale was used to assess patients' average daily pain. The subject rated his/her average pain from 0 (no pain) to 10 (worst pain ever experienced).
  The average pain experienced in the last 7 days was calculated by the mean of the daily Likert Pain Scores within the 7 days prior to the respective visit (ie, Likert Pain Scores with a date of assessment before the date of visit and on or after the date of visit - 7 days). A negative value indicates an improvement.
Time Frame: Baseline (Visit 2) until End of the Maintenance Period (Maintenance Period lasts 12 weeks ± 5 days after an up to 7 weeks Titration Period)
Population: The Analysis Population refers to the Full Analysis Set (FAS). The FAS is a subset of the Safety Set and includes all subjects who were randomized, received at least 1 dose of study medication, and had a valid primary efficacy Baseline measurement and at least 1 valid post-Baseline Maintenance or valid Withdrawal primary efficacy measurement.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 30 | 30
scores on a scale | -2.2 (2.78) | -2.8 (1.84)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.172, ANCOVA; ANCOVA model for the change from Baseline to the End of Treatment containing treatment and region as factors and Baseline value as a covariate; Least Square Mean = -0.76, 95% CI 2-sided [-1.87 to 0.34], Standard Error of Mean 0.55

2. Secondary Outcome: Percentage of Responders at the End of the Maintenance Period
Description: Responders are defined as patients experiencing a 2-Point or more Reduction on an 11-Point Likert Pain Scale from Baseline to the End of the Maintenance Period. An 11-Point Likert Scale was used to assess patients' average daily pain. The patient rated his/her average pain from 0 (no pain) to 10 (worst pain ever experienced).
Time Frame: Baseline (Visit 2) until End of the Maintenance Period (Maintenance Period lasts 12 weeks ± 5 days after up to 7 weeks Titration Period)
Population: as for outcome 1
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 30 | 30
percentage of responders | 46.7 | 60

3. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the Sum Score of the 8-Item Parkinson's Disease Questionnaire (PDQ-8)
Description: The 8-Item Parkinson's Disease Questionnaire (PDQ-8) (Peto et al, 1998) is a self-administered questionnaire that provides a reliable measure of overall health status. The PDQ-8 contains 8 items of daily living, with 1 item selected from each of the following 8 scales: mobility, Activities of Daily Living (ADL), emotional well being, stigma, social support, cognitions, communication, and bodily discomfort. The total PDQ-8 score is the sum of all the individual items converted to a summary index score between 0 and 100, with lower scores indicating better health. A negative value indicates an improvement.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 30
scores on a scale | -3.77 (13.93) | -12.40 (19.25)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.038, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -8.01, 95% CI 2-sided [-15.56 to -0.46], Standard Error of Mean 3.77

4. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the 7-Item Depression Subscore of the Hospital Anxiety and Depression Scale (HADS)
Description: The Hospital Anxiety and Depression Scale (HADS) (Zigmond and Snaith, 1983) is a 14-item self-assessment scale for detecting states of depression and anxiety in the setting of a hospital medical outpatient clinic. It comprises a 7-item anxiety subscale and a 7-item depressive subscale that are also measures of severity of the emotional disorder. The 14 items are scored between 0 and 3. The 7-item depression subscore and 7-item anxiety subscore were calculated as the sum of the 7 corresponding individual scores. A negative value indicates an improvement.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 28 | 28
scores on a scale | -1.7 (4.3) | -1.9 (4.1)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.247, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -1.02, 95% CI 2-sided [-2.76 to 0.73], Standard Error of Mean 0.87

5. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the 7-Item Anxiety Subscore of the Hospital Anxiety and Depression Scale (HADS)
Description: as for outcome 4
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 28 | 28
scores on a scale | -1.0 (3.2) | -1.8 (3.7)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.371, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -0.58, 95% CI 2-sided [-1.85 to 0.70], Standard Error of Mean 0.64

6. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the Combined Score of the Unified Parkinson's Disease Rating Scale (UPDRS) Parts II (Activities of Daily Living [ADL] Subscale) and III (Motor Subscale)
Description: Part II of the Unified Parkinson's Disease Rating Scale (UPDRS) assesses the subject's activities of daily living. Part III assesses motor function. The UPDRS is completed by questioning the subject about his/her general state in conjunction with any observations made by the investigator (or designee) since the previous visit. Part II is subject-rated and Part III is physician-rated. The UPDRS Part II (Activities of Daily Living) consists of 13 items scored between 0 and 4. The sum score was calculated as the sum of these 13 individual scores. The UPDRS Part III (motor subscale) consists of 27 items and sub items scored between 0 and 4. The sum score was calculated as sum of these 27 individual scores. The sum score of UPDRS Parts II and III is the sum of the corresponding single sum scores. A negative value indicates an improvement.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 30
scores on a scale | -5.1 (11.7) | -8.3 (11.2)
Statistical Analysis 1: Comparison: Placebo vs Rotigotine; Test type: Superiority or Other; p = 0.346, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Square Mean = -2.82, 95% CI 2-sided [-8.76 to 3.13], Standard Error of Mean 2.97

7. Secondary Outcome: Change From Baseline to the End of the Maintenance Period in the 7 Domain Scores of Classification of Pain in Parkinson's Disease
Description: The classification of pain in Parkinson's disease scale classifies pain in the following domains: musculoskeletal pain (item 1), chronic pain (items 2 and 3), fluctuation related pain (items 4, 5 and 6), nocturnal pain (items 7 and 8), oro-facial pain (items 9, 10 and 11), discoloration; edema/swelling (items 12 and 13), and radicular pain (item 14). Severity of the pain is measured on a scale from none (0) to severe (3) and frequency is measured on a scale from never (0) to very frequent (4).
  A score of a single item was calculated by multiplying severity with frequency. A domain score was calculated as the sum of every individual score related to the respective domain. A negative value indicates an improvement.
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Rotigotine
Number analyzed (Participants) | 29 | 30
scores on a scale
  Musculoskeletal Pain | -1.4 (3.6) | -1.5 (4.2)
  Chronic Pain | -3.1 (5.6) | -0.7 (2.9)
  Fluctuation-Related Pain | -2.2 (4.6) | -4.2 (6.8)
  Nocturnal Pain | -2.9 (6.1) | -2.4 (5.3)
  Oro-Facial Pain | -0.4 (2.5) | -0.6 (2.3)
  Discoloration; Edema/Swelling | -1.8 (4.9) | -1.7 (3.4)
  Radicular Pain | -1.3 (3.8) | -1.1 (3.7)

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events were reported from Baseline up to the Safety Follow-up Visit (approximately during 25 weeks).
Description: Adverse Events refer to the Safety Set (SS). The SS includes all randomized subjects who received at least 1 dose of study medication.
Arm/Group | Placebo | Rotigotine
Serious Adverse Events (participants affected / at risk) | 1/33 | 2/35
Other Adverse Events (participants affected / at risk) | 17/33 | 20/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=33) | Rotigotine (N=35)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=33) | Rotigotine (N=35)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 8 (11)
Application site erythema (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Dyskinesia (Nervous system disorders) | 2 (2) | 2 (2)
Hyperkinesia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 4 (11) | 6 (7)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days